CLINICAL TRIAL: NCT02232789
Title: Abuse Liability and Human Pharmacology of Mephedrone (4-methylmethcathinone,4-MMC)
Brief Title: Abuse Liability and Human Pharmacology of Mephedrone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: IMIMFTCL/MEF/1
Record Dates: First submitted 2014-08-29; First posted 2014-09-05 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Amphetamine-Related Disorders
Keywords: Mephedrone; 3,4-methylenedioxymethamphetamine; Abuse liability; Human Pharmacology
MeSH Terms: conditions — Amphetamine-Related Disorders | interventions — mephedrone; N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mephedrone (Experimental): Mephedrone 200 mg, single dose, oral administration
  Interventions: Drug: Mephedrone
- 3,4-methylenedioxymethamphetamine (Active Comparator): 3,4-methylenedioxymethamphetamine (MDMA) 100 mg, single dose, oral administration
  Interventions: Drug: 3,4-methylenedioxymethamphetamine
- Lactose (Placebo Comparator): Placebo, single dose, oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mephedrone — Single oral dose mephedrone
  Other Names: 4-methylmethcathinone; 4-MMC
  Arms: Mephedrone
Drug: 3,4-methylenedioxymethamphetamine — Single oral dose MDMA
  Other Names: MDMA; Ecstasy
  Arms: 3,4-methylenedioxymethamphetamine
Drug: Placebo — Single oal dose placebo
  Other Names: Non active treatment
  Arms: Lactose

SUMMARY:
The purposes of this study are 1) to evaluate the abuse liability and human pharmacology of mephedrone after oral administration and 2) to compare the pharmacological effects of mephedrone with those obtained after administration of oral 3,4-methylenedioxymethamphetamine (MDMA, ecstasy).

DETAILED DESCRIPTION:
Mephedrone is a new psychoactive substance (NPS). At present, there are no randomized controlled trials evaluating the effects of mephedrone in humans. The current body of knowledge regarding the acute effects of mephedrone is based on anecdotal, self-reported effects (e.g. internet forums), case reports, and emergency room series and fatalities.

The aims of this study are 1) to evaluate the abuse liability and human pharmacology of mephedrone after oral administration and 2) to compare the pharmacological effects of mephedrone with those obtained after administration of oral 3,4-methylenedioxymethamphetamine (MDMA, ecstasy).

ELIGIBILITY:
Inclusion Criteria:

* Understanding and accepting the study procedures and signing the informed consent.
* Male adults volunteers (18-45 years old).
* Clinical history and physical examination demonstrating no organic or psychiatric disorders.
* The ECG and general blood and urine laboratory tests performed before the study should be within normal ranges. Minor or occasional changes from normal ranges are accepted if, in the investigator's opinion, considering the current state of the art, they are not clinically significant, are not life-threatening for the subjects and do not interfere with the product assessment. These changes and their non-relevance will be justified in writing specifically.
* Recreational use of amphetamines, ecstasy and hallucinogen derivatives, mephedrone or other cathinone on at least 6 occasions (two in the previous year) without serious adverse reactions.
* Extensive metabolizer or intermediate metabolizer phenotype for cytochrome P-450-2D6 (CYP2D6) activity determined using dextromethorphan as a selective probe drug.
* The weight does not exceed 15% of ideal weight that applies according to size and will be between 60 and 100 Kg. Minor variations will be accepted as normal limits, if the researchers considered it clinically insignificant.

Exclusion Criteria:.

* Daily consumption >20 cigarettes and >4 standard units of ethanol.
* Regular use of any drug in the month prior to the study sessions. The treatment with single or limited doses of symptomatic medicinal products in the week prior to the study sessions will not be a reason for exclusion if it is calculated that it has been cleared completely the day of the experimental session.
* Presence of major psychiatric disorders.
* Present history of abuse or drug dependence (except for nicotine dependence).
* Past history of drug dependence (except for nicotine dependence). Subjects with past history of drug abuse could be included.
* Having suffered any organic disease or major surgery in the three months prior to the study start.
* Blood donation 12 weeks before or participation in other clinical trials with drugs in the previous 4 weeks.
* Subjects with intolerance or serious adverse reactions to drugs or amphetamines, ecstasy and hallucinogen derivatives, mephedrone or other cathinone.
* History or clinical evidence of gastrointestinal, liver, renal or other disorders which may lead to suspecting a disorder in drug absorption, distribution, metabolism or excretion, or that suggest gastrointestinal irritation due to drugs.
* Subjects unable to understand the nature, consequences of the study and the procedures requested to be followed.
* Subjects with positive serology to Hepatitis B, C or HIV.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Changes in blood pressure | From pre-dose (baseline) to 4h post-dose
  Systolic and diastolic blood pressure

SECONDARY OUTCOMES:
Changes in euphoria-good effects | From pre-dose (baseline) to 4h post-dose
  Euphoria-good effects effects will be measured using rating scales (visual analogue scales, the Addiction Research Center Inventory and the Evaluation of the Subjective Effects of Substances with Abuse Potential questionnaires). All these instruments include measures of euphoria-good effects and other feelings induced by psychostimulants
Area Under the Concentration-Time Curve (AUC 0-24h) | From baseline (pre-dose, 0h) to 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 24h post-dose
  Calculation of AUC of the concentrations of mephedrone and MDMA and its metabolites in blood, urine, oral fluid and sweat.
Number of Participants with Serious and Non-Serious Adverse Events | 7 days after each substance administration
  Collection of adverse effects spontaneously reported by the participants and/or observed by the investigators
Elimination half-life | From baseline to 24h post-dose
  Calculation of elimination hal-life from concentrations of mephedrone, MDMA and its metabolites in plasma-blood, urine, oral fluid and sweat.
Changes in heart rate | From pre-dose (baseline) to 4h post-dose
  Measure of heart rate (pulse)
Changes in pupil diameter | From pre-dose (baseline) to 4h post-dose
  Measure of pupil diameter and capacity of convergence (esophoria) using a pupillometer
Changes in oral temperature | From pre-dose (baseline) to 4h post-dose
  Measure of temperature in mouth using automatic thermometer

CONTACTS AND LOCATIONS:
Overall Officials: Magi Farre, MD, PhD, Principal Investigator — Parc de Salut Mar
Locations (1):
- Institut Hospital del Mar d'Investigacions Mèdiques-IMIM. Parc de Salut Mar., Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Papaseit E, Perez-Mana C, Mateus JA, Pujadas M, Fonseca F, Torrens M, Olesti E, de la Torre R, Farre M. Human Pharmacology of Mephedrone in Comparison with MDMA. Neuropsychopharmacology. 2016 Oct;41(11):2704-13. doi: 10.1038/npp.2016.75. Epub 2016 May 20. PMID 27206266